CLINICAL TRIAL: NCT06903650
Title: Evaluation of the Effect of Salpingectomy Operation on Ovarian Reserve With Anti-Mullerian Hormone and Ovarian Doppler Ultrasonography
Brief Title: The Effect of Salpingectomy Operation on Ovarian Reserve
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Derya Öztürk, Principal Investigator, Dokuz Eylul University
Other Study IDs: SOORAMHODU
Record Dates: First submitted 2025-03-21; First posted 2025-03-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Insufficiency
Keywords: Salpingectomy; Ovarian Reserve; Anti-Mullerian Hormone; Doppler Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- perioperative ovarian arter pulsatility index(PI)(right and left), perioperative AMH levels
  Interventions: Procedure: bilateral salpingectomy, ovarian arter doppler ultrasonography
- postoperative days 2 ovarian arter pulsatility index (PI) (right and left)
  Interventions: Procedure: bilateral salpingectomy, ovarian arter doppler ultrasonography
- postop. weeks 6 ovarian arter pulsatility index(PI)(right and left), postop. weeks 6 AMH levels
  Interventions: Procedure: bilateral salpingectomy, ovarian arter doppler ultrasonography

INTERVENTIONS:
Procedure: bilateral salpingectomy, ovarian arter doppler ultrasonography — The effect of salpingectomy operation on ovarian reserve

SUMMARY:
This study aimed to evaluate the effect of salpingectomy operation on ovarian reserve. Ovarian reserve was evaluated by measuring anti-mullerian hormone levels from serum samples taken from the patients before the operation and 6 weeks after the operation. Ovarian doppler flow were evaluated by measuring the ovarian artery pulsatility index with transvaginal ultrasonography preoperatively, postoperative days 2 and postoperative weeks 6 . In our study, it was determined that ovarian functions may be negatively affected in the acute period after salpingectomy operation.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 37-45 with continuing menstrual cycles (37 and 45 included)
2. Patients who will undergo uterine surgery for benign reasons or who will undergo salpingectomy only due to hydrosalpinx, ectopic pregnancy, tubo-ovarian abscess
3. Patients who have not had ovarian surgery before
4. Those without menopause and premature ovarian failure
5. Patients who accept the study

Exclusion Criteria:

1. Age younger than 37 or older than 45
2. Those who want to withdraw from the study
3. Those who do not come for follow-up examination
4. Use of drugs that affect ovarian reserve
5. Any surgical procedure performed on the ovaries during the operation
6. No menstrual bleeding in the last year
7. Patients who received radiotherapy and hormonal therapy within 3 months before surgery

Ages: 37 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Serum samples will be separated from routine blood samples taken from patients who apply to the outpatient clinic and will undergo salpingectomy within the indication, during perioperative preparation and at the 6th week postoperatively, after patient consent is obtained. This serum sample will be taken into an Eppendorf tube and kept at -40˚C for later AMH levels to be studied. Ovarian artery pulsatility index values measured during the patient's perioperative and postoperative routine ultrasonographic examination and weeks 6 postoperative control will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
right ovarian arter pı | perioperative, postoperative days 2 , postoperative weeks 6
  rate of 0,87/ 0,84/ 0,76
left ovarian arter pı | perioperative, postoperative days 2, postoperative weeks 6
  rate of 0,89/ 0,79/ 0.80
AMH levels | perioperative-postoperative weeks 6
  Concentration of 1 ng/mL / 0,79 ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No